CLINICAL TRIAL: NCT06261970
Title: Leveraging and Strengthening Local Systems to Increase First-time Mothers' Use of Postpartum Family Planning in Tanzania: A Cluster Randomized Control Trial
Brief Title: Increase First-time Mothers' Use of Postpartum Family Planning in Tanzania: The Connect Project
Acronym: Connect TZ
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: George Washington University (Other)
Collaborators: Save the Children (Other); Save the Children International Tanzania (Unknown); Bill and Melinda Gates Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 999002684
Record Dates: First submitted 2024-02-08; First posted 2024-02-15 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Contraceptive Usage
MeSH Terms: conditions — Contraception Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Connect Community Level Enhancements (Experimental): Community Support Groups (CSGs)*: Connect enhances Lishe Endelevu's to require at least four FTMs to be recruited into each CSG established. Connect enhances the CSG toolkit to include FTM focused content, including information on birth spacing and PPFP.
  Home visits*: the CHWs who facilitate the community support groups also conduct home visits to FTMs. CHWs are provided a job aid to counsel FTMs and their families on PPFP. Counseling addresses myths about FP, norms around fertility and spacing, and includes prompts to engage family and male partners when present. Counseling also integrates timely nutrition information from the support groups with PPFP information. CHWs can provide non-clinical FP methods (pills, condoms) and provide referrals for services at public health facilities
  Interventions: Behavioral: Connect
- Control (No Intervention): No additional Connect intervention. Lishe Endelevu Community Support Groups Operate per usual.

INTERVENTIONS:
Behavioral: Connect — Community level enhancements
  Arms: Connect Community Level Enhancements

SUMMARY:
While a growing body of programs have shown promise to increase use of contraception among first time mothers (FTMs), difficulties remain in scaling beyond small pilot areas and institutionalizing within existing systems. Connect's approach aims to strengthen existing government health systems and community-level health efforts, including those supported through local and international non-governmental organizations, by developing and testing light-touch "enhancements" with the goal of increasing postpartum Family Planning (PPFP) adoption among FTMs. The investigators will evaluate Connect's approach through a cluster randomized control trial.

DETAILED DESCRIPTION:
While a growing body of programs have shown promise to increase use of contraception among first time mothers (FTMs), difficulties remain in scaling beyond small pilot areas and institutionalizing within existing systems. Connect's approach aims to strengthen existing government health systems and community-level health efforts, including those supported through local and international non-governmental organizations, by developing and testing light-touch "enhancements" with the goal of increasing postpartum Family Planning (PPFP) adoption among FTMs. The investigators will evaluate Connect's approach through a cluster randomized control trial.

The overall goal of this study is to add to the evidence base on scalable and efficacious approaches for increasing PPFP uptake among adolescent and young FTMs in order to increase spacing before subsequent births and improve maternal and neonatal outcomes.

Specifically, this protocol outlines the parameters for the evaluation of the impact of Connect's package of interventions-or "enhancements"-on adoption and continued use of modern PPFP methods among adolescent (ages 15-19 years) and young (ages 20-24 years) FTMs. These interventions are community support groups (CSGs) with PPFP-specific content and enhanced training for community health workers (CHWs) around PPFP for delivery during home visits.

Alongside the wider-scale implementation of these enhancements, Connect will support the Ministry of Health as well as local and international non governmental organizations (NGOs) to sustain the enhancements beyond the donor-funded project.

There are four specific aims for understanding the efficacy for Connects packages:

1. To estimate the causal impact and cost-effectiveness of Connect's community-level interventions (compared to a control) on the primary outcomes of adoption and continuation of modern PPFP methods among FTMs ages 15-24 in two districts in Tanzania.
2. To examine the causal impact of Connect's community-level interventions (compared to a control) on secondary outcomes (specified below) among FTMs ages15-24 in two districts in Tanzania.
3. To compare the impacts of Connect's community-level interventions on adolescent FTMs (ages 15-19) versus young FTMs (ages 20-24).
4. To use mixed-methods research to unpack the mechanisms by which the various interventions work, as well as understand for whom they work and why (exploratory analysis).

ELIGIBILITY:
Inclusion Criteria:

* Pregnant or has child under 9 months
* Aged 14-25

Exclusion Criteria:

* Younger than 14 or over 25
* Has more than one child or is pregnant and has a child

Ages: 14 Years to 25 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Gender Based: Yes — Self identifies as first time mother
Enrollment: 1134 (Actual)
Dates: Start 2023-02-22 (Actual); Primary Completion 2025-02-02 (Actual); Study Completion 2025-02-02 (Actual)

PRIMARY OUTCOMES:
Adoption of of Postpartum Family Planning (PPFP): | 12 months
  1. Indicator for adopted a modern contraceptive method within 12 months after giving birth (among women who have given birth). Adoption of a modern contraceptive method in the first year after giving birth, among FTMs who have given birth-modern methods are defined here as male condoms, oral contraceptive pills, injectables, and long-active reversible contraception (LARC) methods (implants and intrauterine device (IUD)). We will use the following indicators to measure adoption and continuation of PPFP:
Currently Using PPFP | At time of 12 month survey
  Currently using a modern contraceptive method (among women who have given birth). modern methods are defined here as male condoms, oral contraceptive pills, injectables, and long-active reversible contraception (LARC) methods (implants and intrauterine device (IUD)).

SECONDARY OUTCOMES:
Adopted or Intention to adopt PPFP | 12 months
  1. Indicator for adopt or intention to adopt modern PPFP with 12 months after birth
  * Using or planning to use a modern contraceptive method to delay or avoid pregnancy within first year of child's life, among all FTMs who have given birth within the past 12 months
  * Modern methods included in this indicator are: male condoms, oral contraceptive pills, injectables, implants, IUDs
Average Satisfaction with PPFP methods | 12 months
  2. Indicator for FTM believes advantages outweigh disadvantages, average across methods used, among those who have given birth
  o Methods: male condom, pill, injectable, implant, IUD
Contraceptive Preferences | 12 Months
  3. Contraceptive preferences for modern methods, among all FTMs
  o Indicator equal to one if the FTM names a modern method (male condom, pill, injectable, implant, IUD) as preferred family planning method if there were no constraints (e.g., cost, access, opinions of others, etc.).
Quality of Family Planning Counseling | 12 months
  Quality score (0-100), among all FTMs who received family planning counseling A 22-item quality of care index, adapted from Jain et al. (2019) is combined into a weighted additive index where each of 4 domains have equal weight (1) respectful care, (2) method selection, (3) effective use of method selected, and (4) continuity of contraceptive use and care. For each domain, we will construct an indicator equal to one of the care is of "high quality", defined as having a score that is greater than the mean score plus half of the standard deviation
Communication and Agency | 12 months
  5. Indicator for FTM discussed FP with husband/partner or other family member, among all FTMs
PPFP Attitudes | 12 months
  PPFP attitudes index of nine attitudes, standardized to the mean and standard deviation of the control group, among all FTMs. The raw index will be the sum of the responses to each individual attitude (score ranging from 1 to 5), with a possible maximum score of 45. Higher scores will indicate less restrictive attitudes with regard to family planning.
  o A set of 9 questions using a 5-point likert scale (1=strongly agree, 5=strongly disagree) adapted from EMERGE and PMA 2020 asked in a random order: o
PPFP Knowledge | 12 months
  PPFP knowledge index of eight true/false statements, standardized to the mean and standard deviation of the control group, among all FTMs. The raw index will be the sum of the responses to each individual true/false statement. Raw scores range from 0 to 8, with 8 indicating that all questions were answered correctly.

CONTACTS AND LOCATIONS:
Overall Officials: Sarah Baird, PhD, Principal Investigator — George Washington University
Locations (2):
- Tanzania (2):
  - EDI, Bahi, Dodoma
  - EDI, Kongwa, Dodoma

IPD SHARING:
Plan to Share IPD: Yes
Deidentified data will be made publicly available
Supporting Information: Study Protocol, SAP
Time Frame: 2025